CLINICAL TRIAL: NCT03850210
Title: The Manchester Short Splint in the Rehabilitation of Zone II Flexor Tendon Repairs
Acronym: Short Splint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2015BP001
Record Dates: First submitted 2019-02-13; First posted 2019-02-21 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Tendon Injuries
MeSH Terms: conditions — Tendon Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Splint (Experimental)
  Interventions: Device: Short Splint
- Traditional, Long Splint (Active Comparator)
  Interventions: Device: Traditional Long Splint

INTERVENTIONS:
Device: Short Splint — Short Splint that permits maximal wrist flexion and up to 45° of wrist extension with a block to 30° of MCP joint extension.
  Arms: Short Splint
Device: Traditional Long Splint — Traditional splint is a forearm-based dorsal thermoplastic splint that immobilizes the wrist in neutral position with a block to 30° of metacarpophalangeal (MCP) joint extension
  Arms: Traditional, Long Splint

SUMMARY:
The project sets out to compare two different splints in the outcome of zone II flexor tendon injury hand therapy rehabilitation programme. Traditional hand therapy is based on using a long forearm-based splint for 6 weeks in zone II flexor tendon injuries. Manchester University NHS Foundation Trust have devised a new shorter splint to use as an alternative to the traditional longer splint as there are cogent reasons for believing that permitting more wrist movement during rehabilitation will improve the range of finger movement ultimately (tendonesis effects).

Patients will be randomised to receive either the traditional long splint, or the short splint. Patients will be followed up and data will be collected at routine hand therapy appointments.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients 16 years and over, undergoing surgical repair of zone II flexor tendon injury in a single digit

Exclusion Criteria:

* Adult patients lacking capacity or motivation to participate in the planned physiotherapy
* Adult patients with special needs and vulnerable groups
* Adult patients who undergo surgical repair of their flexor tendon more than 4 days after the initial injury
* Patients unable to understand English adequately
* Adult patients unable to attend the hospital facility for the requisite number of planned physiotherapy sessions (social reasons)
* Adult patients with multiple level injuries
* Injuries with soft tissue loss requiring coverage
* Adult patients with two nerve injuries on the same finger
* Adult patients with multiple digit flexor tendon injury
* Adult patients with concomitant bony injury to the hand
* Children under 16 years age

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in range of motion of the proximal interphalangeal joint of the injured digit at baseline and 6 months | Active and passive motion ranges to be recorded at 3 and 6 months
  Range of motion of the proximal interphalangeal joint of the injured digit as measured by hand therapist using goniometer (angle measuring device)

SECONDARY OUTCOMES:
Rupture of repaired flexor tendon | Monitored at 3 and 6 months
  • Rupture of repaired flexor tendon which is assessed and determined clinically by the treating hand therapist and confirmed by the responsible surgeon. Determined ruptured when there is no 'pull through' and the finger does not flex on attempted active movement
Tendon adhesions needing tenolysis | Monitored at 3 and 6 months
  • Tendon adhesions diagnosed by differential active/passive range of motion as measured by hand therapist using goniometer. Confirmed by responsible surgeon

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No